CLINICAL TRIAL: NCT00610311
Title: Phase II Study of Metastatic Melanoma Using Lymphodepleting Conditioning Followed by Infusion of Anti-gp100:154-162 TCR-Gene Engineered Lymphocytes and ALVAC Virus Immunization
Brief Title: Anti-gp100 Cells Plus ALVAC gp100 Vaccine to Treat Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to low accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080055; 08-C-0055
Record Dates: First submitted 2008-02-06; First posted 2008-02-07 (Estimated); Results first posted 2012-04-10 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-09

CONDITIONS: Metastatic Melanoma; Skin Cancer
Keywords: Metastatic Melanoma; Immunotherapy; Vaccination; Tumor Regression; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Cyclophosphamide; fludarabine phosphate; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALVAC plus anti-gp100:154-162 TCR PBL + HD IL-2 (Experimental): ALVAC plus anti-gp100:154-162 T cell receptor (TCR) peripheral blood lymphocytes (PBL) + high dose (HD) interleukin-2 (IL-2): ALVAC vaccine two hours prior to cell infusion patients will receive 0.5 ml containing a target dose of 10^7 cell culture infectious dose 50% (CCID50) (with a range of approximately 10^6.4 to 107.9/mL of the gp100 ALVAC virus subcutaneously in each extremity (total of 4 x 10^7 CCID50/2mL. This will be repeated on day 14.
  Aldesleukin (IL2, Proleukin, Recombinant human interleukin 2)- 720,000 IU/kg intravenous over 15 minutes every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses)
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Biological: Aldesleukin; Biological: ALVAC gp100 Vaccine; Biological: anti-gp100:154-162 Tcell receptor (TCR) peripheral blood lymphocyte (PBL)

INTERVENTIONS:
Drug: cyclophosphamide — 60 mg/kg day x 2 days intravenous in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg day x 2 days over 1 hour
  Other Names: Cytoxan
Drug: fludarabine phosphate — 25 mg/m^2 day intravenous piggy back over 30 minutes for 5 days
  Other Names: Fludara
Biological: Aldesleukin — 720,000 IU/kg intravenously over 15 minutes every 8 hours (+/- 1 hour) for up to 5 days.
  Other Names: Proleukin
Biological: ALVAC gp100 Vaccine — 0.5 ml containing a target dose of 10^7 CCID50 (with a range of approximately 10^6,4 to 10^7,9/mL) of the gp100 ALVAC virus subcutaneously in each extremity (total of 4 x 10^7 CCID50/2mL)
  Other Names: ALVAC
Biological: anti-gp100:154-162 Tcell receptor (TCR) peripheral blood lymphocyte (PBL) — 3 x 10^11 anti-gp100:154-162 TCR engineered PBL by intravenous infusion. A minimum of approximately 5 x 10^8 cells will be given.

SUMMARY:
Background:

* gp100 is a protein that is often found in melanoma tumors.
* An experimental procedure developed for treating patients with melanoma uses anti-gp100 cells designed to destroy their tumors. The anti-gp100 cells are created in the laboratory using the patient's own tumor cells or blood cells.
* The treatment procedure also uses a vaccine called plaque purified canarypox vector (ALVAC) gp100, made from a virus that ordinarily infects canaries and is modified to carry a copy of the gp100 gene. The virus cannot reproduce in mammals, so it cannot cause disease in humans. When the vaccine is injected into a patient, it stimulates cells in the immune system that may increase the efficiency of the anti gp 100 cells.

Objectives:

-To evaluate the safety and effectiveness of anti-gp100 cells and the ALVAC gp100 vaccine in treating patients with advanced melanoma.

Eligibility:

-Patients with metastatic melanoma for whom standard treatments have not been effective.

Design:

* Patients undergo scans, x-rays and other tests and leukapheresis to obtain white cells for laboratory treatment.
* Patients have 7 days of chemotherapy to prepare the immune system for receiving the gp100 cells.
* Patients receive the ALVAC vaccine, anti-gp100 cells and interleukin-2 (IL-2) (an approved treatment for advanced melanoma). The anti gp100 cells are given as an infusion through a vein. The vaccine is given as injections just before the infusion of gp100 cells and again 2 weeks later. IL-2 is given as a 15-minute infusion every 8 hours for up to 5 days after the cell infusion for a maximum of 15 doses.
* After hospital discharge, patients return to the clinic for periodic follow-up with a physical examination, review of treatment side effects, laboratory tests and scans every 1 to 6 months.

DETAILED DESCRIPTION:
Background:

* We have engineered human peripheral blood lymphocytes (PBLs) to express a T-cell receptor that recognizes an human leukocyte antigens (HLAA) 0201 restricted epitope derived from the gp100 protein.
* We constructed a single retroviral vector that contains both alpha and infinity chains and can mediate genetic transfer of this T cell receptor (TCR) with high efficiency (greater than 30 percent) without the need to perform any selection.
* In co-cultures with HLA-A 0201 positive melanoma gp100:154-162 TCR transduced T cells secreted significant amount of interferon (IFN)-(but no significant secretion was observed in control co-cultures with cell lines.

gp100:154-162 TCR transduced PBL could efficiently kill -HLA-A 0201 positive tumors. There was little or no recognition of normal fibroblasts cells.

* This TCR is over 10 times more reactive with melanoma cells than the melanoma antigen recognized by T-cells (MART)-1 TCR that mediated tumor regression in two patients with metastatic melanoma.
* In this trial we would like to test our hypothesis that the addition of an anti-tumor ALVAC vaccine will result in clinical tumor regression, and persistence of the transferred cells (as is the case in murine models).

Objectives:

Primary objectives:

-Determine if the administration of anti-gp100:154-162 TCR-engineered peripheral blood lymphocytes, ALVAC anti-tumor immunization, and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic melanoma.

Secondary objectives:

* Determine the in vivo survival of TCR gene-engineered cells.
* Determine the toxicity profile of this treatment regimen.
* Determine whether treated patients develop anti-mouse TCR antibody.

Eligibility:

Patients who are HLA-A 0201 positive and 18 years of age or older must have:

* metastatic melanoma;
* previously received and have been a non-responder to or recurred after aldesleukin;
* normal values for basic laboratory values.

Patients may not have:

* concurrent major medical illnesses;
* any form of primary or secondary immunodeficiency;
* severe hypersensitivity to any of the agents used in this study;
* contraindications for high dose aldesleukin administration.

Design:

* Peripheral blood mononuclear cells (PBMC) obtained by leukapheresis (approximately 5 times 10^9 cells) will be cultured in the presence of anti-CD3 (OKT3) and aldesleukin in order to stimulate T-cell growth.
* Transduction is initiated by exposure of approximately 10^8 to 5 times 10^8 cells to supernatant containing the anti-gp100:154-162 TCR retroviral vector. These transduced cells will be expanded and tested for their anti-tumor activity.
* Once engineered PBMC are demonstrated to be biologically active according to the strict criteria outlined in the Certificate of Analysis, patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of ex vivo tumor reactive, TCR gene-transduced PBMC plus intravenous (IV) aldesleukin (720,000 IU/kg q8h for a maximum of 15 doses). Approximately 2 hours prior to cell infusion, patients will be immunized with ALVAC virus expressing the tumor antigen. ALVAC immunization will be repeated at 2 weeks.
* Patients will undergo complete evaluation of tumor with physical examination, computed tomography (CT) of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment and then monthly for approximately 3 to 4 months or until off study criteria are met.
* The study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled. If 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled.
* The objective will be to determine if the combination of high dose aldesleukin, lymphocyte depleting chemotherapy, ALVAC immunization and anti-gp100:154-162 TCR-gene engineered lymphocytes is able to be associated with a clinical response rate that can rule out 5 percent (p0=0.05) in favor of a modest 20 percent partial response (PR) plus complete response (CR) rate (p1=0.20).

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Metastatic melanoma with measurable disease.
2. Previously received high dose interleukin-2 (IL-2) and have been either non-responders (progressive disease) or have recurred.
3. Positive for gp100 by immunohistochemistry (IHC) which will be reviewed by the Laboratory of Pathology at National Cancer Institute (NCI).
4. Tumor infiltrating lymphocyte (TIL) cells not available for treatment on other Surgery Branch protocols.
5. Greater than or equal to 18 years of age.
6. Willing to sign a durable power of attorney.
7. Able to understand and sign the Informed Consent Document.
8. Clinical performance status of Eastern Oncology Oncology Group (ECOG) 0 or 1.
9. Life expectancy of greater than three months.
10. Patients of both genders must be willing to practice birth control for four months after receiving the preparative regimen.
11. Must be human leukocyte antigens (HLA-A) 0201 positive.
12. Serology:

    * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol-depends on an intact immune system. Patients who are HIV seropositive can have decreased immune -competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative.
13. Hematology:

    * Absolute neutrophil count greater than 1000/mm^3.
    * White blood cell (WBC) (greater than 3000/mm^3).
    * Platelet count greater than 100,000/mm^3.
    * Hemoglobin greater than 8.0 g/dl.
14. Chemistry

    * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to 2.5 times the upper limit of normal.
    * Serum creatinine less than or equal to 1.6 mg/dl.
    * Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
15. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
16. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
17. Six weeks must have elapsed since prior MDX-010 therapy to allow antibody levels to decline, and patients who have previously received MDX-010 or ticilimumab must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
2. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Ongoing opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
5. Systemic steroid therapy.
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. History of coronary revascularization.
8. Documented left ventricular ejection fraction (LVEF) of less than 45 percent in patients with:

   * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, 2 degree or 3 degree heart block.
   * Age greater than or equal to 60 years old.
9. Documented forced expiratory volume in 1 second (FEV1) less than or equal to 60 percent predicted for patients with:

   * A prolonged history of cigarette smoking (greater than 20 pack/year within the past 2 years).
   * Symptoms of respiratory distress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Rivoltini L, Topalian SL, Miki T, Rosenberg SA. Cloning of the gene coding for a shared human melanoma antigen recognized by autologous T cells infiltrating into tumor. Proc Natl Acad Sci U S A. 1994 Apr 26;91(9):3515-9. doi: 10.1073/pnas.91.9.3515. PMID 8170938
- [Background] Kawakami Y, Eliyahu S, Sakaguchi K, Robbins PF, Rivoltini L, Yannelli JR, Appella E, Rosenberg SA. Identification of the immunodominant peptides of the MART-1 human melanoma antigen recognized by the majority of HLA-A2-restricted tumor infiltrating lymphocytes. J Exp Med. 1994 Jul 1;180(1):347-52. doi: 10.1084/jem.180.1.347. PMID 7516411
- [Background] Walter EA, Greenberg PD, Gilbert MJ, Finch RJ, Watanabe KS, Thomas ED, Riddell SR. Reconstitution of cellular immunity against cytomegalovirus in recipients of allogeneic bone marrow by transfer of T-cell clones from the donor. N Engl J Med. 1995 Oct 19;333(16):1038-44. doi: 10.1056/NEJM199510193331603. PMID 7675046
- See also: Response Evaluation Criteria in Solid Tumors (RECIST) Criteria — http://ctep.cancer.gov/protocolDevelopment/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three participants was enrolled in this study.
Groups:
- ALVAC Plus Anti-gp100:154-162 TCR PBL + HD IL-2: ALVAC plus anti-gp100:154-162 T cell receptor (TCR) peripheral blood lymphocytes (PBL) + HD interleukin-2 (IL-2): ALVAC vaccine two hours prior to cell infusion patients will receive 0.5 ml containing a target dose of 10^7 CCID50 (with a range of approximately 10^6.4 to 107.9/mL of the gp100 ALVAC virus subcutaneously in each extremity (total of 4 x 10^7 CCID50/2mL. This will be repeated on day 14.
  3 x 10^11 anti-gp100:154-162 TCR engineered PBL by intravenous infusion. A minimum of approximately 5 x 10^8 cells will be given.
  Aldesleukin (IL2, Proleukin, Recombinant human interleukin 2)- 720,000 IU/kg intravenous over 15 minutes every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses)
Period: Overall Study
Arm/Group | ALVAC Plus Anti-gp100:154-162 TCR PBL + HD IL-2
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ALVAC Plus Anti-gp100:154-162 TCR PBL + HD IL-2
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Metastatic Melanoma Who Develop Clinical Tumor Regression (CR or PR)
Description: Clinical tumor response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v.1.0 criteria. Complete response (CR) is a disappearance of all target lesions. Partial response (PR) is a 30% decrease in lesions taking as reference the baseline sum longest diameter (LD). For details about the RECIST criteria see the protocol link module.
Time Frame: 4-6 weeks after treatment and then monthly for approximately 3 to 4 months or until off study criteria are met
Measure: Number; unit: Participants
Arm/Group | ALVAC Plus Anti-gp100:154-162 TCR PBL + HD IL-2
Number analyzed (Participants) | 3
Participants
  Partial response (PR) | 1
  Complete response (CR) | 0

2. Secondary Outcome: Number of Participants With in Vivo Survival of T-cell Receptor (TCR) Gene-engineered Cells.
Description: T cell receptor (TCR) and vector presence will be quantitated in peripheral blood mononuclear cells (PBMC) samples using established polymerase chain reaction (PCR) techniques. This will provide data to estimate the in vivo survival of lymphocytes derived from the infused cells.
Time Frame: 1 month
Population: This outcome measure was not done because the study was terminated due to low accrual.
Arm/Group | ALVAC Plus Anti-gp100:154-162 TCR PBL + HD IL-2
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 18.5 months
Measure: Number; unit: Participants
Arm/Group | ALVAC Plus Anti-gp100:154-162 TCR PBL + HD IL-2
Number analyzed (Participants) | 3
Participants | 3

4. Secondary Outcome: Number of Participants Who Develop Anti-mouse T Cell Receptor (TCR) Antibodies
Description: Blood samples are collected from the patient and an immunological test is conducted in the laboratory to determine if the patient has generated antibodies against the mouse T-cell receptor which is part of the anti-gp100 cells.
Time Frame: 1 month
Population: This outcome measure was not done because the study was terminated due to low accrual.
Arm/Group | ALVAC Plus Anti-gp100:154-162 TCR PBL + HD IL-2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 18.5 months
Groups:
- ALVAC Plus Anti-gp100:154-162 TCR PBL + HD IL-2: ALVAC plus anti-gp100:154-162 T cell receptor (TCR) peripheral blood lymphocytes (PBL) + HD interleukin-2 (IL-2): ALVAC vaccine two hours prior to cell infusion patients will receive 0.5 ml containing a target dose of 10^7 CCID50 (with a range of approximately 10^6.4 to 107.9/mL of the gp100 ALVAC virus subcutaneously in each extremity (total of 4 x 10^7 CCID50/2mL. This will be repeated on day 14.
  Aldesleukin (IL2, Proleukin, Recombinant human interleukin 2)- 720,000 IU/kg intravenous over 15 minutes every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses)
Arm/Group | ALVAC Plus Anti-gp100:154-162 TCR PBL + HD IL-2
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALVAC Plus Anti-gp100:154-162 TCR PBL + HD IL-2 (N=3)
Intracranial hemorrhage (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALVAC Plus Anti-gp100:154-162 TCR PBL + HD IL-2 (N=3)
Hearing test abnormal (Ear and labyrinth disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2)
Leukocyte count decreased (Blood and lymphatic system disorders) | 3 (3)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 3 (3)
Neutrophil count decreased (Blood and lymphatic system disorders) | 3 (4)
Platelet count decreased (Blood and lymphatic system disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Activated partial thromboplastin time prolonged (aPTT) (Investigations) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 3 (3)
Creatinine increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (3)
Uveitis (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Low urine output (Renal and urinary disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No